CLINICAL TRIAL: NCT04256863
Title: Examining the Role of Chrononutrition in Behavioral Weight Control for Adolescents
Brief Title: Chrononutrition and Adolescent Weight Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202819; U54GM115677 (NIH)
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-01

CONDITIONS: Adolescent Obesity; Diet; Weight Loss; Sleep
MeSH Terms: conditions — Pediatric Obesity; Weight Loss | interventions — Breakfast; Lunch; Meals

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast / Lunch (BFL) (Experimental): This group will complete a 16-week standard behavioral weight control intervention in which they will be asked to consume >50% of their daily energy goal before 3PM. To do so, they will complete weekly experiential learning sessions in conjunction with the SBT lessons.
  Interventions: Behavioral: Breakfast / Lunch
- Dinner (DIN) (Active Comparator): This group will complete a 16-week standard behavioral weight control intervention. They will not be given any recommendations regarding the timing of their energy consumption, but instead encouraged to follow the same energy goals at the BFL group.
  Interventions: Behavioral: Dinner (DIN)

INTERVENTIONS:
Behavioral: Breakfast / Lunch — Participants in the BFL group will participate in 16 weekly, group based sessions weekly sessions in which they will be exposed to standard behavioral therapy (SBT) for weight control. Each 90-minute session will cover one weight control topic (self-monitoring, modifying the home food environment, physical activity, goal setting, stimulus control, stress-related eating, motivation, problem solving, healthy eating on a budget, social influences and weight loss maintenance) and an experiential learning activity. These hands-on activities will help teens build skills to adhere to 1) their calorie goal (1,400 - 1,600 calories/day) and 2) the prescribed timing for consumption (>50% of their energy needs consumed before 3PM every day of the week. Sample meal plans will be provided to help with adherence. .
  Arms: Breakfast / Lunch (BFL)
Behavioral: Dinner (DIN) — Participants randomized to the Dinner (DIN) group will participate in the same 16-week intervention as those in the BFL group; however, the topics covered in the experiential learning session will pertain to skills needed to adhere to prescribed calorie goals NOT to timing. They will be instructed to consume >50% of their energy needs after 3PM daily.; however, given that most teens consume the bulk of their calories after 5PM, the focus will be on general calorie goals vs. timing., Teens in this group will also be provided sample meal plans that outline how to spread out their calorie intake across breakfast (200), lunch (300), after school snack (200 calories), Dinner (700 calories), after dinner snack (200 calories for 1,600 calorie diet only).
  Arms: Dinner (DIN)

SUMMARY:
Comprehensive lifestyle interventions are recommended for the treatment of adolescent obesity; however, evidence suggests that they are not as effective in teens as they are in children and adults. Recent evidence supports that shifting the timing of energy intake earlier in the day has led to improved weight loss outcomes among adults with overweight and obesity. Given that adolescents traditionally consume the majority of their daily energy intake late in the day (past 5PM), this approach may improve the effectiveness of traditional behavioral weight control interventions in teens. Therefore, the primary aim of the proposed research is to pilot a novel adaptation of an evidence-based adolescent weight control intervention in which adolescents will be randomized to consume the majority of their daily energy needs earlier versus later in the day. More specifically, 40 adolescents, ages 13-17, with obesity (BMI>95% for age and sex) will be randomized to a 16-week evidence-based weight control intervention that has the participant consume >50 percent of their total energy intake before 3PM (i.e. at breakfast / lunch; BFL) or after 3PM (i.e. dinner; DIN). Assessments will take place at baseline and 16 weeks (post-treatment). The proposed study will test 1) the adherence and feasibility of the BFL vs. DIN interventions as measured by the average number of days on which daily energy was consumed in accordance with the prescribed eating plan and, secondarily, mean session attendance, 2) if the BFL group will have significantly greater reductions in BMI post-treatment as compared to the DIN group, 3) if there are differences in sleep duration and quality between groups, and finally, as an exploratory aim, whether there are differences in dietary quality between groups. The proposed research is significant, as it addresses obesity in teens. It is innovative as the timing of meals and snacks have not been manipulated in adolescents in the context of behavioral weight control. Moreover, the study will shed light on whether doing so improves sleep and could help to untangle how sleep and weight gain relate in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age 13- 17 years
* BMI > 85th percentile for age and sex
* Ability to speak, read and write English due to the group format of the intervention
* A caregiver who is willing to participate in four separate parent groups with a facilitator
* Agreement to study participation and random assignment.

Exclusion Criteria:

* Current involvement in another weight loss program or has lost 10 pounds in the six months prior to enrollment
* Medical condition that interferes with the prescribed dietary plan or participation in physical activity (e.g. cardiovascular disease, type 1 or 2 diabetes mellitus, or pregnancy)
* In treatment for or are diagnosed with a major psychiatric disorder, including an eating disorder, at the time of screening
* Taking medications that promote weight gain.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility: Percent of energy consumed | 3 weeks (mid-intervention)
  Percent of energy consumed before 3PM (BFL) or after 3PM (DIN) will be measured using data from weekly diet records from weeks 8, 9, and 10. During these three weeks, the interventionist will determine the number of days that each participant consumed >50% of their daily calories in accordance with their prescribed eating plan (before 3PM (BFL) or after 3PM (DIN)). Thus, each participant will receive a score out of total possible 21 days.
Adherence | 16-week intervention
  Participant attendance in weekly group-based sessions

SECONDARY OUTCOMES:
Change in Body Mass Index z-score (BMIz) | Baseline and Immediately after intervention (16 weeks)
  Change in BMIz, which will be calculated based on height and weight measurements collected at baseline and 16-weeks (end of intervention) assessments
Change in Sleep Duration | Baseline and Immediately after intervention (16 weeks)
  Participants will wear actigraphs and complete a sleep-log at baseline and at the end of the intervention to measure sleep duration, which is the number of minutes between sleep onset and rise time scored sleep.
Change in Sleep Quality: proportion of the sleep period spent asleep and not awake | Baseline and Immediately after intervention (16 weeks)
  Participants will wear actigraphs and complete a sleep-log at baseline and at the end of the intervention to measure sleep quality, which is defined as the proportion of the sleep period spent asleep and not awake

CONTACTS AND LOCATIONS:
Overall Officials: Erin W Evans, PhD, Principal Investigator — The Miriam Hospital; Jared Saletin, PhD, Principal Investigator — The Bradley Hospital
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States